CLINICAL TRIAL: NCT01221753
Title: A Phase II Study of Docetaxel/Cisplatin/5-Fluorouracil (TPF) Induction Chemotherapy Followed by Concurrent Chemoradiotherapy Using a Modified Radiation Dose in Patients With Newly Diagnosed HPV Positive, Locally Advanced Squamous Cell Carcinoma of the Oropharynx
Brief Title: Docetaxel/Cisplatin/5-Fluorouracil (TPF) Human Papillomavirus (HPV) Squamous Cell Carcinoma Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to slow accrual
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Robert I. Haddad, MD, Medical Oncology, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-038
Record Dates: First submitted 2010-09-21; First posted 2010-10-15 (Estimated); Results first posted 2016-12-06 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-11

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck; Human Papilloma Virus
Keywords: SSCHN; HPV; IMRT
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Docetaxel; Cisplatin; Fluorouracil; Radiotherapy, Intensity-Modulated; Cetuximab; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TPF Induction Chemotherapy followed by Chemoradiotherapy (Experimental): Patients received 3 cycles (21 days each) of TPF induction chemotherapy: docetaxel 75 mg/m2 IV day 1; cisplatin 100 mg/m2 IV day 1 (carboplatin substitute permitted); 5-FU 1000 mg/m2/day IV pump continuous days 1-4. Concurrent chemoradiotherapy followed 4-6 weeks after day 1 of cycle 3 TPF induction: cetuximab 400 mg/m2 IV loading dose 1 week prior and 250 mg/m2 IV weekly (panitumumab substitute permitted); carboplatin AUC 1.5 (Calvert formula) IV weekly; Intensity modulated radiation therapy (IMRT)-response based dosing for 6-7 weeks.
  Interventions: Drug: docetaxel; Drug: cisplatin; Drug: 5-FU; Radiation: IMRT; Drug: cetuximab; Drug: carboplatin

INTERVENTIONS:
Drug: docetaxel
  Other Names: Taxotere; Docefrez
Drug: cisplatin — Given intravenously on day 1 of each cycle
  Other Names: Platinol-AQ
Drug: 5-FU
  Other Names: 5-fluorouracil
Radiation: IMRT
  Other Names: Intensity modulated radiation therapy
Drug: cetuximab
  Other Names: Erbitux
Drug: carboplatin
  Other Names: Paraplatin

SUMMARY:
In this research study, the investigators are studying whether a reduced dose of radiation when given with standard doses of chemotherapy can reduce side effects without compromising control of the cancer. An approved treatment for squamous cell carcinoma of the head and neck is initial chemotherapy followed by radiation and chemotherapy together. This treatment is effective but has many immediate and long-term side effects. People who have squamous cell carcinoma of the head and neck (SSCHN) that is related to an infection by the human papillomavirus (HPV) have been shown to have a high response to this treatment along with a high cure rate. The investigators think that by reducing the intensity of this treatment, they may be able to reduce immediate and long-term side effects which may lead to long term improvements in quality of life and function.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

To determine rate of local-regional control at 2 years

Secondary

To determine Progression Free Survival at 2 and 5 years

To determine Overall Survival at 2 and 5 years

To assess acute toxicity and long term toxicity of reduced radiation dose at 2 and 5 years

ELIGIBILITY:
Inclusion Criteria

* Histologically or cytologically confirmed squamous cell carcinoma of the oropharynx or unknown primary that is HPV 16 positive as determined by ISH and p16 positive as determined by IHC.
* Stage 3 or 4 disease without evidence of distant metastases
* At least one evaluable or uni- or bi-dimensionally measurable lesion by RECIST 1.1 criteria
* 18 years of age or older
* No previous surgery, radiation therapy or chemotherapy for SSCHN is allowed at time of study entry
* ECOG Performance Status of 0 or 1
* No active alcohol addiction
* Adequate bone marrow, hepatic and renal function as defined in the protocol
* Women of child-bearing potential must have a negative pregnancy test within 7 days of starting treatment

Exclusion Criteria

* Pregnant or breast feeding women or women and men of childbearing potential not willing to use adequate contraception while on treatment and for at least 3 months after
* Previous or current malignancies at other sites
* Symptomatic peripheral neuropathy of grade 2 or greater
* Symptomatic altered hearing greater than grade 2
* Other serious illnesses or medical conditions
* Patients that have experienced an involuntary weight loss of more than 25% of their body weight in the 2 months preceding study entry
* Concurrent treatment with any other anticancer therapy
* Participation in an investigational trial within 30 days of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-07; Primary Completion 2012-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Haddad, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is no data available.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 7 participants were enrolled between July 2011 and May 2012.
Period: Overall Study
Arm/Group | TPF Induction Chemotherapy Followed by Chemoradiotherapy
Started | 7
Completed | 6
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | TPF Induction Chemotherapy Followed by Chemoradiotherapy
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: 2-Year Local-Regional Control Rate
Description: 2-year local-regional control rate is defined as the proportion of participants who achieve confirmed stable disease (SD) or better by 2-years post study registration based on RECIST 1.0 criteria. Per RECIST 1.0 for target lesions, complete response (CR) is disappearance of all target lesions and partial response (PR) is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. Progressive disease (PD) is at least a 20% increase in sum LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started. SD is neither PR nor PD. For non-target lesions, PD is the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: Follow-up for response continued until first progression. Disease assessments occurred at completion of induction cycle 3 along with months 12, 18 and 24 post study registration.
Population: The study was terminated early due to weak accrual. Clinical outcome data were not accessible for results reporting due to the designation of study completed at the institution.
Arm/Group | TPF Induction Chemotherapy Followed by Chemoradiotherapy
Number analyzed (Participants) | 0

2. Secondary Outcome: 4-y Overall Survival Rate
Description: 4-year overall survival rate is the percentage of patients remaining alive 4-years from study entry.
Time Frame: Patients were followed for survival up to 5 years from study entry. Patients alive have been followed for a mean of 55 months (range 52-60 months).
Population: The analysis dataset is comprised of all treated patients. Since all patients have not been followed for survival for 5 years the 4-year rate is provided. All data provided was based on chart review and not from case report forms.
Measure: Number; unit: percentage of participants
Arm/Group | TPF Induction Chemotherapy Followed by Chemoradiotherapy
Number analyzed (Participants) | 7
percentage of participants | 100

ADVERSE EVENTS:
Time Frame: Assessed each cycle throughout induction, weekly during chemoradiotherapy and until outstanding adverse events are stable or resolved. All patients completed treatment (3 cycles of TPF induction and 7 weeks of chemoradiotherapy). AEs with treatment-attribution of possibly, probably or definitely were classified as serious if maximum grade 3-5 or other if grade 1-2 per CTCAEv4.There is no accessible AE data at this point.
Description: The study was terminated early due to weak accrual. AE data were not accessible for results reporting due to the designation of study completed at the institution conduction the study.
Arm/Group | TPF Induction Chemotherapy Followed by Chemoradiotherapy
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The study was terminated early due to weak accrual. Because of the designation of study completed at the institution conducting the study, data collected systematically on the case report forms were not accessible for results reporting.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes